CLINICAL TRIAL: NCT06426589
Title: Resistance Training and Mediterranean Diet in the Mental Health of the Older Adult Population: a Randomized Controlled Clinical Trial
Brief Title: Exercise and Nutrition in the Mental Health of the Older Adult Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Responsible Party: Principal Investigator, Agustín Aibar Almazán, Principal investigator, University of Jaén
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UJA.2024
Record Dates: First submitted 2024-05-17; First posted 2024-05-23 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Older Adults
MeSH Terms: interventions — Diet, Mediterranean

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): The control group (CG) will not undergo treatment, which will be evaluated in the pre- and post-phase of the study. Participants assigned to this group will receive general advice on the positive effects of regular physical activity, and they will be given the guide of recommendations for the promotion of physical activity.
- Experimental Group (Experimental): The experimental group (EG), after an initial evaluation, will be subjected to a physical training program based on the resistance training, for 12 weeks with 2 weekly sessions (Tuesday and Thursday), with a duration of 45 minutes per session. Once the intervention is finished, you will undergo a final evaluation again to see if there is a difference or not with the results obtained at the beginning. In addition to the resistance training intervention, the experimental group received a Mediterranean diet protocol.
  Interventions: Other: Resistence training and mediterranean diet

INTERVENTIONS:
Other: Resistence training and mediterranean diet — Resistance training. Subjects assigned to the experimental group participated in resistance program twice a week (on Tuesdays and Thursdays) for a period of 12 weeks, totaling 24 sessions of 60 minutes each. Each session during this time was divided into three clearly differentiated parts: i) 5-minute warm-up comprised of a series of gentle, low-intensity exercises designed to gradually prepare the muscles and joints of older adults for the main exercise.
  Mediterranean Diet. In addition to the resistance intervention, the experimental group received a Mediterranean diet protocol based on the study by Ismail et al. [34] with the following meal plan: i) carbohydrates constituted 50% of daily intake; ii) fats repre-sented 35%; and iii) proteins accounted for 15%.
  Arms: Experimental Group

SUMMARY:
Resistance exercise and the Mediterranean diet are complementary, evidence-based approaches to improving physical and mental health throughout all stages of life.

For older adults, maintain flexibility, muscle strength, balance and posture, reducing the risk of falls and injuries; They relieve chronic pain, improve sleep quality, and reduce stress and anxiety. For young people, they improve concentration, attention and memory, reduce stress and anxiety, promote a positive body image and increase self-esteem. Overall benefits include promoting the mind-body connection, facilitating healthy aging, and being accessible and adaptable to various individual and socioeconomic needs.

The main components of the Mediterranean diet are: high in fruits, vegetables, legumes, nuts, whole grains, fish and olive oil; moderate in dairy and red wine; and low in red meat and processed products. Benefits for older adults include reducing the risk of cardiovascular disease, decreasing chronic diseases and pro-inflammatory factors, and preventing obesity and cognitive decline. The overall impact improves bone and cardiovascular health, and strengthens the immune system.

The combination of resistance exercise and a Mediterranean diet offers a comprehensive approach to improving health and well-being throughout life, promoting physical and mental health, facilitating active and healthy aging, and being accessible and beneficial for people of all socioeconomic backgrounds

ELIGIBILITY:
Inclusion Criteria:

* Were 65 years or older were eligible for the study
* Had not been part of any resistance program in the last 12 months
* They could understand and follow the instructions, activities and protocols of the exercise program.

Exclusion Criteria:

* They suffered from any systemic condition (e.g., neurodegenerative, musculoskeletal, or visual diseases) that prevented them from performing the exercises.
* Had any vestibular disease or disorder
* Consumed medications that influenced the central nervous system, balance or coordination (for example, antidepressants, vestibular sedatives or anxiolytics).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 108 (Actual)
Dates: Start 2023-10-23 (Actual); Primary Completion 2024-01-19 (Actual); Study Completion 2024-01-26 (Actual)

PRIMARY OUTCOMES:
Adherence to the Mediterranean Diet | Up to twelve weeks
  This was measured using the 14-item Mediterranean Diet Adherence Questionnaire (MEDAS) questionnaire, developed by the Prevention with Mediterranean Diet (PREDIMED) researchers. The questionnaire consists of 12 queries regarding how often various foods are eaten and two additional questions concerning typical eating habits in Spain [35]. Each question could be answered with a score of either zero or one. The total possible score ranged from 0 to 14, with a total of 9 or higher signifying sufficient compliance with the Mediterranean diet.
Anxiety and depression | Up to twelve weeks
  To evaluate anxiety and depression levels, the Hospital Anxiety and Depression Scale (HADS) was used [36,37]. This instrument is frequently used in populations of older adults who are not institutionalized [38] and includes 14 questions, divided equally between anxiety (even questions) and depression (even questions). Items are scored on a scale of 0 to 3, resulting in a total score range of 0 to 21 for both anxiety and depression, with a higher number indicating a greater presence of symptoms.
  Sleep quality
Sleep quality | Up to twelve weeks
  The Pittsburgh Sleep Quality Index (PSQI) [39,40], a widely recognized tool for the assessment of sleep quality, was the questionnaire selected for this task. The PSQI includes 19 self-report items and 5 additional items that must be completed by the participant's bed partner or roommate (the latter are used only to obtain clinical data). From these items, a global score is calculated and seven dimensions or areas are evaluated: sleep quality; time to fall asleep; sleep duration; sleep efficiency; problems during sleep; consumption of sleep medication; and daytime functioning problems. The total score on the PSQI ranges from 0 to 21, with higher scores indicating poor sleep quality.
Perceived stress | Up to twelve weeks
  The measurement of perceived stress was carried out using the Perceived Stress Scale (PSS) [41] in its version for the Spanish language [42], an instrument composed of 14 questions that determines the degree of stress felt in the last month. This questionnaire uses a response system based on a five-point scale (0 = never, 1 = almost never, 2 = occasionally, 3 = frequently, 4 = very frequently). To calculate the total score on the PSS, the response values for items 4, 5, 6, 7, 9, 10, and 13 are reversed (so that 0 becomes 4, 1 becomes 3, etc.) and Then all the items are added. The score ranges from 0-56, with a higher score on the scale indicating a higher level of perceived stress.

CONTACTS AND LOCATIONS:
Locations (1):
- Agustín Aibar Almazán, Jaén, Spain

IPD SHARING:
Plan to Share IPD: No